CLINICAL TRIAL: NCT06635044
Title: Effect of Intradialytic Exercise on Erectile Dysfunction in Hemodialysis Men
Acronym: IDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Mohamed Mazen (Other)
Collaborators: Delta University for Science and Technology (Other)
Responsible Party: Sponsor-Investigator, Mohammed Mohamed Mazen, lecturer of physical therapy, Delta University for Science and Technology
Organization: Delta University for Science and Technology (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F.P.T2407028
Record Dates: First submitted 2024-08-28; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IDEP group (Experimental): a pedal exerciser (RTL10273 Deluxe Folding Pedal Exerciser, Drive Medical Co. MPN) was utilized in performing leg cycling exercises while men were sitting. Before starting the session of intradialytic cycling, a 5-minute stretching of the lower limbs was performed as a warming up. Also, as cooling down, the same period of lower limbs' stretching was performed after ending intradialytic cycling
  Interventions: Other: intradialytic exercise
- control group (No Intervention): this group served as waitlist men.

INTERVENTIONS:
Other: intradialytic exercise — HD men came to the HD unit three times weekly to receive their dialysis session which consumed 3-4 hours. During the first two hours of the men's dialysis session, a pedal exerciser (RTL10273 Deluxe Folding Pedal Exerciser, Drive Medical Co. MPN) was utilized in performing leg cycling exercises while men were sitting. Before starting the session of intradialytic cycling, a 5-minute stretching of the lower limbs was performed as a warming up. Also, as cooling down, the same period of lower limbs' stretching was performed after ending intradialytic cycling
  Arms: IDEP group

SUMMARY:
This study aimed to assess the effect of IDEP on ED and its associated psychological burden in HD men. Forty HD men with ED were randomly assigned into the IDEP group (this group contained 20 HD men with ED who received intradialytic cycling three times per week) and the control group (this group served as waitlist men). outcomes : Five-Item International Index of Erectile Function (FI-IIEF), ten-question Rosenberg self-esteem scale (TQ-RSES), version three of the Revised UCLA Loneliness Scale (LS), the revised version of Impact of Event Scale (RV-IES), Beck's Depression Inventory (BDI), and State-Trait Anxiety Inventory (S-TAI) were assessed before and after 12 weeks.

DETAILED DESCRIPTION:
This study aimed to assess the effect of IDEP on ED and its associated psychological burden in HD men. Forty HD men with ED were randomly assigned into the IDEP group (this group contained 20 HD men with ED who received intradialytic cycling three times per week) and the control group (this group served as waitlist men). outcomes :Five-Item International Index of Erectile Function (FI-IIEF), ten-question Rosenberg self-esteem scale (TQ-RSES), version three of the Revised UCLA Loneliness Scale (LS), the revised version of Impact of Event Scale (RV-IES), Beck's Depression Inventory (BDI), and State-Trait Anxiety Inventory (S-TAI) were assessed before and after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men gender
* Hemodialysis for at least 6 months their
* Age between 35 to 48 years old.
* Married patient
* Education level.
* The problem of ED was diagnosed by a physician at least 6 months before enrollment in this study.

Exclusion Criteria:

* prostatic disorders
* systemic diseases (diabetes mellitus or hypertension)
* cardiac diseases
* musculoskeletal issues (e.g. muscle contusion, osteoarthritis, osteoporosis, osteopenia, etc.),
* persistent hyperkalemia
* penile shaft problems/implants
* malignancies, acute/chronic infection or inflammation
* autoimmune disease
* cerebrovascular accidents/insults
* a history of frequent hypoglycaemic episodes,
* absolute contraindications to cardiopulmonary training/exertion
* respiratory or liver diseases
* participation in another structured interdialytic or intradialytic exercise programs
* neurological diseases
* consumptions of ED pharmacotherapies
* previous pelvic surgeries
* radiotherapy
* low levels of testosterone or sex hormones,
* psychological diseases
* Present history of smoking or alcohol consumption.

Ages: 35 Years to 48 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Five-item international index of erectile function | 12 weeks
  A hard copy of FI-IIEF was given to every HD man with ED to fill it before and after the IDEP.

SECONDARY OUTCOMES:
ten-question Rosenberg self-esteem scale (TQ-RSES), | 12 weeks
  ten questions/statements. Four-point Likert responses were allocated to every question/statement of the ten-question Rosenberg self-esteem scale (TQ-RSES).

OTHER OUTCOMES:
version three of the Revised UCLA Loneliness Scale (LS), | 12 weeks
  This scale was used to assess HD patients' loneliness. Four-point Likert responses were allocated to every question/statement of this 20-item scale.
the revised version of Impact of Event Scale (RV-IES), | 12 weeks
  The RV-IES tool/questionnaire is commonly utilized in clinical trials to monitor subjects' stress to recent and/or specific traumatic events. Five-point Likert responses were allocated to every question/statement of this 22-item scale
Beck's Depression Inventory (BDI) | 12 weeks
  This inventory was used to assess depression in this study's participants. The assessed HD patients' BDI contained 21 questions/items
State-Trait Anxiety Inventory (S-TAI) | 12 weeks
  S-TAI is a psychologically self-reported valid/reliable inventory/questionnaire used to examine two main forms of anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Rehan Abdelaziz, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No